CLINICAL TRIAL: NCT02239692
Title: A Randomised, Assessor-blinded, Multi-centre Trial Comparing the Efficacy, Safety and Tolerability of the PICOPREP Tailored Dosing Schedule to the PICOPREP Day-before Dosing Schedule for Colon Cleansing in Preparation for Colonoscopy
Brief Title: A Trial Comparing the PICOPREP Tailored Dosing Schedule to the PICOPREP Day-before Dosing Schedule for Colon Cleansing in Preparation for Colonoscopy
Acronym: OPTIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 000121; 2014-001062-10 (EudraCT Number)
Record Dates: First submitted 2014-09-09; First posted 2014-09-15 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Bowel Cleansing
MeSH Terms: interventions — picosulfate sodium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICOPREP day-before dosing schedule (Active Comparator): Both doses administered the day before colonoscopy.
  Interventions: Drug: PICOPREP
- PICOPREP tailored dosing schedule (Experimental): First dose one day before colonoscopy or on the day of colonoscopy, dependent on the planned time for colonoscopy, and second dose on the day of colonoscopy.
  Interventions: Drug: PICOPREP

INTERVENTIONS:
Drug: PICOPREP — Sodium Picosulfate, Magnesium Oxide and Citric Acid as PICOPREP powder for oral solution

SUMMARY:
This was a phase 3, randomised, assessor-blinded, multi-centre trial comparing the efficacy, safety and tolerability of a PICOPREP tailored dosing schedule to the PICOPREP day-before dosing schedule for colon cleansing in preparation for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or above, being scheduled to undergo elective colonoscopy
* Subjects must have had more than or equal to 3 spontaneous bowel movements (i.e. without use of any laxative within 24 hours before the bowel movement, with the exception for bulk-forming laxatives (ATC code A06AC)) per week for one month prior to the colonoscopy

Exclusion Criteria:

* Acute surgical abdominal conditions (e.g. acute obstruction or perforation, etc.)
* Active (acute/exacerbation of/severe/uncontrolled) Inflammatory Bowel Disease (IBD)
* Any prior colorectal surgery, excluding appendectomy, haemorrhoid surgery or prior endoscopic procedures
* Colon disease (history of colonic cancer, toxic megacolon, toxic colitis, idiopathic pseudoobstruction, hypomotility syndrome)
* Ascites
* Gastrointestinal disorder (active ulcer, outlet obstruction, retention, gastroparesis, ileus)
* Upper gastrointestinal surgery (gastric resection, gastric banding, gastric by-pass)
* Severely reduced renal function (Glomerular filtration rate (GFR) <30 (mL/min/1.73 m2))
* The subject is a pregnant (positive urine pregnancy test at Visit 1 or Visit 2) woman. Women of childbearing potential (defined, for the purpose of this trial, as all females post-puberty, not postmenopausal ≥2 years, or not surgically sterile) who do not agree to use one of the following methods of birth control from the day of signing the Informed Consent Form until End of Trial Visit are excluded:

  1. Transdermal patch
  2. Hormonal contraception (i.e., oral, implant, or injectable contraceptive)
  3. Double-barrier birth control (i.e., condom plus intrauterine device, diaphragm plus spermicide, etc.)
  4. Maintenance of a monogamous relationship with a male who has been surgically sterilised by vasectomy
  5. Sexual abstinence
* The subject is a breast-feeding or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (3):
- Ed Herriot Hopital (there may be other sites in this country), Lyon, France
- Gastroenterologie am Bayerischen Platz (there may be other sites in this country), Berlin, Germany
- Medisch Centrum Alkmaar (there may be other sites in this country), Alkmaar, Netherlands

REFERENCES:
- [Derived] Kiesslich R, Schubert S, Mross M, Klugmann T, Klemt-Kropp M, Behnken I, Bonnaud G, Keulen E, Groenen M, Blaker M, Ponchon T, Landry W, Stoltenberg M. Efficacy and safety of PICOPREP tailored dosing compared with PICOPREP day-before dosing for colon cleansing: a multi-centric randomised study. Endosc Int Open. 2017 Apr;5(4):E282-E290. doi: 10.1055/s-0043-102433. PMID 28393103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11 sites in Germany, France and the Netherlands from Nov 2014 to Jun 2015.
Groups:
- PICOPREP Day-before Dosing Schedule: Dose 1 was given before 8:00 AM on day before colonoscopy and Dose 2 was given 6-8 hours after Dose 1.
  PICOPREP: Sodium Picosulfate, Magnesium Oxide and Citric Acid as PICOPREP powder for oral solution
- PICOPREP Tailored Dosing Schedule: Dose 1 was given 10-18 hours before colonoscopy and Dose 2 was given 4-6 hours before colonoscopy.
  PICOPREP: Sodium Picosulfate, Magnesium Oxide and Citric Acid as PICOPREP powder for oral solution
Period: Overall Study
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Started | 73 | 131
Intention-to-treat Analysis Set | 73 | 131
Per-protocol Analysis Set | 66 | 120
Safety Analysis Set | 70 | 125
Completed | 67 | 118
Not Completed | 6 | 13
Not completed — Incomplete colonoscopy | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Other reason | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) analysis set consisted of all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule | Total
Number analyzed (Participants) | 73 | 131 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 85 | 134
  >=65 years | 24 | 46 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (15.1) | 58.4 (13.3) | 57.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 77 | 120
  Male | 30 | 54 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 71 | 128 | 199
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 73 | 130 | 203
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Colon Cleansing Procedure (ITT) Measured by the Total Ottawa Scale
Description: Measured by the total Ottawa Scale score during the colonoscopy performed by a colonoscopist blinded to the dosing schedules. Total Ottawa Scale score was computed by adding the ratings (0 to 4; 0=excellent, 1=good, 2=fair, 3=poor, 4=inadequate) for each of the three colon segments and the overall fluid quality rating (0 to 2). The final score ranged from 0 (excellent) to 14 (solid stool in each colon segment and lots of fluid).
Time Frame: Day 1 (day of colonoscopy)
Population: The ITT analysis set consisted of all randomized subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Number analyzed (Participants) | 73 | 131
score on a scale | 8.2 (3.54) | 4.2 (3.75)
Statistical Analysis 1: Comparison: PICOPREP Day-before Dosing Schedule vs PICOPREP Tailored Dosing Schedule; Null hypothesis was no treatment difference between the two dosing schedules; Test type: Non-Inferiority or Equivalence — Non-inferiority is assessed by examining whether the upper limit of the 95% confidence interval is less than the specified non-inferiority margin of 1.5 points; p < 0.0001, ANCOVA — p-value corresponds to a two-sided test of superiority; ANCOVA with treatment, country and time of colonoscopy (AM/PM) as factors; Adjusted estimated mean difference = -3.93, 95% CI 2-sided [-4.99 to -2.87] — Treatment difference in mean total Ottawa Scale score was calculated as PICOPREP tailored dosing schedule minus PICOPREP day-before dosing schedule

2. Primary Outcome: Overall Colon Cleansing Procedure (PP) Measured by the Total Ottawa Scale
Description: Measured by the total Ottawa Scale score during the colonoscopy which is performed by a colonoscopist blinded to the dosing schedules. Total Ottawa Scale score was computed by adding the ratings (0 to 4; 0=excellent, 1=good, 2=fair, 3=poor, 4=inadequate) for each of the three colon segments and the overall fluid quality rating (0 to 2). The final score ranged from 0 (excellent) to 14 (solid stool in each colon segment and lots of fluid).
Time Frame: Day 1 (day of colonoscopy)
Population: The per-protocol (PP) analysis set consisted of all the subjects included in ITT analysis set, but excluding subjects with major protocol deviations (18 subjects) that would impact efficacy analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Number analyzed (Participants) | 66 | 120
score on a scale | 8.1 (3.38) | 3.7 (3.14)
Statistical Analysis 1: Comparison: PICOPREP Day-before Dosing Schedule vs PICOPREP Tailored Dosing Schedule; Null hypothesis was no treatment difference between the two dosing schedules; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANCOVA — p-value corresponds to a two-sided test of superiority; ANCOVA with treatment, country and time of colonoscopy (AM/PM) as factors; Adjusted estimated mean difference = -4.38, 95% CI 2-sided [-5.34 to -3.41] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Ascending Colon Cleansing Responder Status (ITT)
Description: Percentage of subjects classified as responders, i.e. Ottawa Scale score of either 0 (excellent) or 1 (good), during colonoscopy performed by a colonoscopist blinded to the dosing schedules.
Time Frame: Day 1 (day of colonoscopy)
Population: The ITT analysis set consisted of all randomized subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Number analyzed (Participants) | 73 | 131
percentage of subjects | 15.1 | 61.1
Statistical Analysis 1: Comparison: PICOPREP Day-before Dosing Schedule vs PICOPREP Tailored Dosing Schedule; Null hypothesis was no treatment difference between the two dosing schedules; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — p-value corresponds to a two-sided test of superiority; Logistic regression with the failure/success status as dependent variable, and treatment, country and timing of colonoscopy as factors; Adjusted estimated odds ratio = 9.18, 95% CI 2-sided [4.36 to 19.32] — The estimated odds ratio compares the odds of being a responder in the PICOPREP tailored dosing schedule vs. the PICOPREP day-before dosing schedule

4. Secondary Outcome: Frequency and Intensity of Adverse Events
Time Frame: From baseline (screening) up to day 10 after colonoscopy
Population: The Safety analysis set consisted of all treated subjects and was analyzed according to the actual treatment received.
Measure: Number; unit: subjects
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Number analyzed (Participants) | 70 | 125
subjects
  Frequency of all adverse events | 4 | 15
  Frequency of mild adverse events | 4 | 12
  Frequency of moderate adverse events | 0 | 2
  Frequency of severe adverse events | 0 | 1

5. Secondary Outcome: Clinically Significant Changes in Vital Signs (Pulse and Blood Pressure)
Description: Mean change from baseline to the end-of-trial was observed for pulse and blood pressure (systolic and diastolic).
Time Frame: From baseline (screening) up to day 10 after colonoscopy (inclusive of assessment at each visit)
Population: The Safety analysis set consisted of all treated subjects and was analyzed according to the actual treatment received.
Measure: Number; unit: subjects
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Number analyzed (Participants) | 70 | 125
subjects
  Clinically significant change in pulse | 0 | 0
  Clinically significant change in blood pressure | 0 | 0

6. Secondary Outcome: Clinically Significant Changes in Laboratory Values (Haematology, Clinical Chemistry, Coagulation and Urinalysis)
Description: Laboratory parameters included routine haematology, clinical chemistry, coagulation and urinalysis. With the exception of urinalysis and urine pregnancy test, which was performed as dip-stick analyses at the trial site, all laboratory tests were analysed by a central laboratory.
Time Frame: From baseline (screening) up to day 10 after colonoscopy (inclusive of assessment at each visit)
Population: The Safety analysis set consisted of all treated subjects and was analyzed according to the actual treatment received.
Measure: Number; unit: subjects
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Number analyzed (Participants) | 70 | 125
subjects
  Clinically significant change in haematology | 0 | 0
  Clinically significant change in clinical chem | 0 | 0
  Clinically significant change in coagulation | 0 | 0
  Clinically significant change in urinalysis | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from baseline till the end-of-trial (10 days after colonoscopy).
Arm/Group | PICOPREP Day-before Dosing Schedule | PICOPREP Tailored Dosing Schedule
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/125
Other Adverse Events (participants affected / at risk) | 4/70 | 14/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICOPREP Day-before Dosing Schedule (N=70) | PICOPREP Tailored Dosing Schedule (N=125)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICOPREP Day-before Dosing Schedule (N=70) | PICOPREP Tailored Dosing Schedule (N=125)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.